CLINICAL TRIAL: NCT07389915
Title: Design and Validation of a Convolutional Neural Network to Predict Difficult Biliary Canulation: a Multicenter Study.
Brief Title: A Convolutional Neural Network for Difficult Biliary Cannulation
Acronym: PRECABIDO2
Status: Not yet recruiting | Type: Observational
Sponsor: University of La Laguna (Other)
Responsible Party: Principal Investigator, Manuel Hernandez-Guerra, MD, MD, PhD, University of La Laguna
Other Study IDs: CNN difficult cannulation
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-05 (Actual); Status verified 2026-01

CONDITIONS: Difficult Biliary Cannulation
Keywords: ERCP; Difficult biliary cannulation; Convolutional neural network; CNN
MeSH Terms: interventions — Cholangiopancreatography, Endoscopic Retrograde

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients undergoing ERCP: Consecutive patients undergoing endoscopic retrograde cholangiopancreatography (ERCP) will be included
  Interventions: Procedure: Endoscopic retrograde cholangiopancreatography (ERCP)

INTERVENTIONS:
Procedure: Endoscopic retrograde cholangiopancreatography (ERCP) — Patients with a clinical indication of Endoscopic retrograde cholangiopancreatography (ERCP) will be included in the study for malignant or benign conditions as in routine clinical practice. Endoscopic and radiological images of the second portion of the duodenum will be captured for each patient. In patients undergoing endoscopic ultrasound (EUS), additional images of the second portion of the duodenum at the level of the pancreatic head and common bile duct (CBD) will be obtained

SUMMARY:
The main purpose of the study is to train a convolutional neural network (CNN) to predict difficult biliary canulation (DBC) following the European Society of Gastrointestinal Endoscopy Society (ESGE). Consecutive patients undergoing an endoscopic retrograde cholangiopancreatography (ERCP) will be included in the study. Several pictures of the second portion of the duodenum including the ampulla will be taken, along with several pictures of the radiological image. Pictures prospectively collected from the study PRECABIDO (NCT06591364), a multicenter study whith the purpose of evaluating the prevalence of difficult biliary cannulation and predictive factors for difficult cannulation and cannulation failure using ESGE criteria were also used for the training of the CNN.

We will also assess:

A validation of the CNN assessing the agreement between ESGE criteria and the CNN prediction.

To design a novel application based on the use of a convolutional neural network (CNN) to detect difficult biliary cannulation.

.

DETAILED DESCRIPTION:
All consecutive patients who meet the inclusion criteria and none of the exclusion criteria will be offered participation in the study. They will be informed by one of the investigators from each center and will sign an informed consent form. A data collection sheet will be completed to record demographic data, the indication for the procedure, and technical variables.

The procedures will be performed by endoscopists with at least 200 ERCPs and more than 5 years of experience. All patients, except in cases of allergy, will receive 1 suppository of indomethacin or diclofenac before the procedure. In cases of allergy, pre-procedure hydration with Ringer's lactate will be administered if there is no contraindication (consider the protocol proposed by the ESGE: 3 mL/kg/hour during ERCP, 20 mL/kg as a bolus after ERCP, and 3 mL/kg/hour for 8 hours post-ERCP). The use of a pancreatic stent should be considered when indicated.

After the procedure, patients will remain hospitalized for at least 24 hours in the hospital. The patient's medical record will be reviewed 7 days after the procedure to check for any adverse effects, and a follow-up phone call will be made to detect any adverse effects.

Initially, a pilot study will be conducted with 600 patients, assessing based on the results-that is, the percentage of patients with difficult cannulation. At the beginning of the examination, at least three endoscopic images and three radiological images of the second portion of the duodenum will be captured for each patient. In patients undergoing endoscopic ultrasound (EUS), three additional images of the second portion of the duodenum at the level of the pancreatic head and common bile duct (CBD) will be obtained.

These images will be labeled as "CBD yes" or "CBD no" according to ESGE criteria, which will serve as the gold standard. Once labeled, the images will be used to train a convolutional neural network (CNN) capable of predicting, just before attempting biliary cannulation, whether it will be a CBD or not.

The prediction of the trained CNN will be able to be combined with the predictive model of difficult biliary cannulation obtaned from the study PRECABIDO NCT06591364 in order to improve the prediction.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Signed informed consent
* Patients indicated for ERCP

Exclusion Criteria:

* INR > 1.5
* Platelets < 50,000/mm³
* Patients with a prior endoscopic sphincterotomy
* Papilla of Vater not accessible via duodenoscope (gastric or duodenal stenosis due to neoplasm) or gastric surgery (Billroth II, Roux-en-Y)
* Known pancreas divisum
* Indication due to pancreatic duct pathology

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All consecutive patients who meet the inclusion criteria and none of the exclusion criteria will be offered participation in the study.
Sampling Method: Non-Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
To train a convolutional neural network to predict difficult biliary canulation | 1 year
  To train a convolutional neural network to predict difficult biliary canulation following the European Society of Gastrointestinal Endoscopy Society (ESGE): Assessment of difficult biliary cannulation defined by ESGE criteria (> 5 minutes duration until cannulation, > 5 cannulation attempts, > 1 passage of the guidewire into the main pancreatic duct). Based on these criteria pictures will be labelled as difficult biliary cannulation or not

SECONDARY OUTCOMES:
A validation of the CNN | 1 year
  A validation of the CNN assessing the agreement between ESGE criteria and the CNN prediction

IPD SHARING:
Plan to Share IPD: No